CLINICAL TRIAL: NCT02529891
Title: Identification of Volatile Organic Compounds in Exhaled Air During Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: LAVOLEX
Status: Terminated | Type: Observational
Why Stopped: Lack of inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Aide à la Recherche Médicale Ondaine et Environs (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1208090; 2012-A01072-41 (Other: ANSM)
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Volatile Organic Compounds; Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD Patients: Patients with COPD, within 48h after hospital admission for exacerbation.
  Interventions: Other: Measurement of VOC in exhaled air
- non-COPD patients: Healthy person of the entourage of COPD patients.
  Interventions: Other: Measurement of VOC in exhaled air

INTERVENTIONS:
Other: Measurement of VOC in exhaled air — Measurement of VOC in exhaled air during 10 min (tidal breathing) with a portable mass spectrometer

SUMMARY:
Exacerbations of the disease are a hallmark of Chronic Obstructive Pulmonary Disease (COPD), affecting the decline of pulmonary function, quality of life and increasing morbidity. The use of validated biomarkers could help to identify the etiology of exacerbation and to prescribe antibiotherapy when indicated.

The analysis of exhaled air allows measuring different volatile organic compounds (VOC) which reflect local or systemic inflammation and oxidative stress. The relationship between the presence of some of these compounds and the exacerbation of COPD has never been studied.

The aim of this study is to identify a cluster of VOC in COPD patients during an acute exacerbation of the disease, compared to a stable condition (3 months after discharge). Investigators also will seek for a relationship between VOC and the etiology of exacerbation (bacterial, viral, inflammatory).

ELIGIBILITY:
Inclusion Criteria of COPD group:

* COPD stages 2 and 3 of GOLD score (30 ≤ forced expiratory volume at one second (FEV1) < 80% of predicted value),
* exacerbation confirmed clinically (increased dyspnea, cough or expectorations > 48 hours)

Inclusion Criteria of non COPD group:

* No smoker (<100 cigarettes/year)

Exclusion Criteria of COPD group:

* Diagnosis of COPD not confirmed.
* Instable clinical status with respiratory failure and indication of mechanical ventilation.
* Bronchodilator treatment changed
* Antibiotic treatment started in the 10 last days before admission

Exclusion Criteria of non COPD group:

* Chronic inflammatory disease
* Any respiratory disease
* Oral corticosteroid treatment during the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with exacerbation of COPD and Healthy volonteers
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Spectrum of VOC measured with a portable mass spectrometer system | Day 1 (within 48 hours after hospital admission for exacerbation of COPD)
  Spectrum of VOC in exhaled air in patients with COPD compared to those of control subjects. It is measured with a portable mass spectrometer system.

SECONDARY OUTCOMES:
Variation in VOC spectrum in COPD patients measured with a portable mass spectrometer system | 3 months after hospital discharge
  Variation in VOC spectrum in COPD patients during exacerbation and in stable condition (3 months later). It is measured with a portable mass spectrometer system.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic COSTES, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France